CLINICAL TRIAL: NCT05125380
Title: Evaluation of an Human Papillomavirus (HPV) Based Screening Algorithm for Low and Middle Income Countries, by Self-sampling in Ethiopia
Brief Title: Cervical Cancer Screening by Self-sampling in a Cohort of Younger Women in Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Collaborators: Addis Ababa University (Other); Armauer Hansen Research Institute, Ethiopia (Other); Adama Hospital Medical College, Ethiopia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: FBKS 2019-6
Record Dates: First submitted 2021-10-07; First posted 2021-11-18 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer; STI; Human Papilloma Virus; Microbiota
Keywords: LMIC Lowe Middle income country; Screening; Vaginal microbiota
MeSH Terms: conditions — Uterine Cervical Neoplasms; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: The whole cohort is offered an HPV self-sample. The HPV high risk positive women gets randomised into two arms VIA or VIA/VILI at the triage step.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- Triage arm for HPV pos women (Active Comparator): HPV positive women
  Interventions: Diagnostic Test: VIA (Visual Inspection with Acetic acid)
- 2- Triage arm for HPV pos women (Experimental): HPV positive women
  Interventions: Diagnostic Test: VIA (Visual Inspection with Acetic acid) and VILI (Visual Inspection with Lugol's Iodine)

INTERVENTIONS:
Diagnostic Test: VIA (Visual Inspection with Acetic acid) and VILI (Visual Inspection with Lugol's Iodine) — A triage test that involved a gynaecological exam that applies acetic acid and then Lugol's iodine on the surface of the external os of the cervix.
  Arms: 2- Triage arm for HPV pos women
Diagnostic Test: VIA (Visual Inspection with Acetic acid) — A triage test that involved a gynaecological exam that applies acetic acid on the surface of the external os of the cervix.
  Arms: 1- Triage arm for HPV pos women

SUMMARY:
The overall purpose of the project is to evaluate an algorithm for an HPV self-sampling based cervical cancer screening algorithm in a mid-size town in Ethiopia that could be applicable for nationwide implementation in low and middle-income countries (LMIC).

Specific aims are the following:

* To evaluate the algorithm using Visual Inspection with Acetic acid (VIA) and VIA together with Lugol's Iodine (VILI) as triage and to use HPV self-sample to follow up those treated and those with persisting HPV.
* To evaluate the prevalence of Chlamydia trachomatis, Neisseria gonorrhoeae and other STIs in the cohort.
* To determine immune response profiles in high-risk HPV-positive women who cleared, persisted, or developed Cervical Intraepithelial Neoplasia 2/3 (CIN).
* To assess how specific cervicovaginal microbiota compositions are associated with HPV infection, cervical dysplasia, and cancer

ELIGIBILITY:
Inclusion Criteria:

* Can give consent, Age above 18

Exclusion Criteria:

* Women who have undergone hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of VIA and VIA/VILI as triage test | 12 weeks
  All HPV pos women will have a cervical biopsy taken

SECONDARY OUTCOMES:
Prevalence of STI other than HPV | 8 weeks
  Chlamydia Trachomatis, Neisseria Gonnorhea, Ureaplasma Urelytikum/Parvum, Trichomonas Vaginalis, Mycoplasma Genitalium/Hominis
Vaginal Microbiota composition | 24 months
  Assessed in HPV high risk pos women at initiation, who persist and who clear their infection

CONTACTS AND LOCATIONS:
Overall Officials: Adane Mihret, PhD, Principal Investigator — Armauer Hansen Research Institute
Locations (1):
- Adama and Geda Health Center, Ādama, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mekuria S, Assiged N, Biazin H, Borgfeldt C, Abebe T, Mihret A, Forslund O, Jerkeman M. Assessing the feasibility of HPV screening for cervical cancer in pregnant women in Ethiopia. Sci Rep. 2025 Aug 28;15(1):31771. doi: 10.1038/s41598-025-15957-y. PMID 40877387
- [Derived] Mekuria SF, Biazin H, Abebe T, Borgfeldt C, Assegid N, Mihret A, Obsi Nemomsa R, Forslund O, Jerkeman M. Comparing visual inspection with acetic acid, with and without Lugol's Iodine for triage of HPV self-sample positive women in Ethiopia: a randomized controlled trial. Int J Gynecol Cancer. 2024 Nov 4;34(11):1691-1697. doi: 10.1136/ijgc-2024-005694. PMID 39362749